CLINICAL TRIAL: NCT00931203
Title: A Phase II Trial of Celecoxib With Preoperative Chemo- Radiation for Locally Advanced Rectal Cancer
Brief Title: Trial of Celecoxib With Preoperative Chemo- Radiation for Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Changhua Christian Hospital (Other); Chi Mei Medical Hospital (Other); Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other); Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2207
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2009-07

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Celecoxib — Celecoxib (400 mg/d) will be continued from day 1 to 65

SUMMARY:
This is a single arm phase II trial with combined celecoxib, tegafur-uracil, folinate and preoperative radiotherapy for patients with locally advanced rectal cancer. The primary end point is pathological complete response (pCR) rate. The secondary endpoints are toxicities of combined celecoxib and chemoradiation, negative resection margin rate, clinical tumor response by magnetic resonance imaging (MRI), sphincter preservation rate, disease-free survival and overall survival.

DETAILED DESCRIPTION:
The primary objective is to determine the pathological complete response (pCR) of combining preoperative tegafur-uracil, folinate, radiation and celecoxib for locally advanced rectal cancer.

The secondary objectives of this study are to determine:

1. Toxicity profile of combining celecoxib, tegafur-uracil, folinate and preoperative radiation for locally advanced rectal cancer.
2. Negative resection margins (circumferential resection margin) rate.
3. Downstaging rate.
4. Sphincter preservation rate
5. Locoregional and distant failure rate.
6. Overall survival

ELIGIBILITY:
Inclusion Criteria:

1. Patients with resectable or potentially resectable adenocarcinoma of the rectum.
2. Clinical stage by Magnetic Resonance Image (MRI) of pelvis, ultrasonography of liver and Chest X ray: AJCC T2 N1-2M0 or T3-4 N0-2M0 (patients who require diverting loop colostomy are eligible). Nuclear medicine study (whole body bone scan or PET scan) can be performed if clinically indicated.
3. Bi-dimensionally measurable disease by MRI, which can be done with pelvic array coil and intrarectal tube.
4. Age greater than 18 years and < 80 years, ECOG performance status < 2
5. Biopsy proven adenocarcinoma, superior margin of the tumor below the L5-S1 spine junction.
6. WBC > 3.5 x109/L, neutrophil count > 1.5x109/L, platelet count > 100x109/L, serum bilirubin < 1.25xULN (upper limit of normal), AST/ALT < 3x ULN, serum creatinine < 1.25xULN.
7. Informed consent signed.

Exclusion Criteria:

1. Distant metastasis, Prior pelvic irradiation, Inflammatory bowel disease, Medical conditions which preclude radical therapy.
2. History of malignancy within five years (except nonmelanoma skin cancer, CIN cervix).
3. Pregnancy.
4. Hypersensitivity to celecoxib, NSAID, sulfonamides or 5-FU.
5. Cardiovascular disease like congestive heart failure, symptomatic coronary artery disease, or myocardiac infarction.
6. History of peptic ulcer disease or NSAID-related gastrointestinal bleeding
7. Use of aspirin, other NSAID or celecoxib in the two weeks prior to study entry.
8. Patients taking warfarin or other anticoagulating medicine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-07; Primary Completion 2012-06 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the pathological complete response (pCR) of combining preoperative tegafur-uracil, folinate, radiation and celecoxib for locally advanced rectal cancer. | 10 weeks

SECONDARY OUTCOMES:
1.Toxicity profile of combining celecoxib, tegafur-uracil, folinate and preoperative radiation for locally advanced rectal cancer. | > 28 weeks
Negative resection margins (circumferential resection margin) rate. | > 28 weeks
Downstaging rate. | > 28 weeks
Sphincter preservation rate. | > 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lin Wei Wang, MD, Principal Investigator — National Health Research of Institutes, Taiwan Cooperative Oncology Group
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan